CLINICAL TRIAL: NCT00302848
Title: The European Active Surveillance Study on OC Prescribing Practice, Benefits and Safety (EURAS)
Brief Title: European Active Surveillance Study (EURAS)
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Juergen Dinger, MD, PhD, Principal Investigator, Berlin Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG 2000_1
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Contraception
Keywords: Venous thromboembolism; Drospirenone
MeSH Terms: conditions — Venous Thromboembolism | interventions — drospirenone; Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Users of Drospirenone (DRSP)
  Interventions: Drug: Drospirenone
- Users of Levonorgestrel (LNG)
  Interventions: Drug: Levonorgestrel
- Users of other oral contraceptives (OCs)
  Interventions: Drug: Other progestin containing oral contraceptive

INTERVENTIONS:
Drug: Drospirenone
  Groups: Users of Drospirenone (DRSP)
Drug: Levonorgestrel
  Groups: Users of Levonorgestrel (LNG)
Drug: Other progestin containing oral contraceptive
  Groups: Users of other oral contraceptives (OCs)

SUMMARY:
EURAS is a multi-national, controlled, prospective, post-marketing, non-intervention cohort study of new users of drospirenone/ethinylestradiol (DRSP/EE), levonorgestrel/ethinylestradiol (LNG/EE) and other oral contraceptives (OCs) under routine conditions of medical practice in seven European countries. Baseline survey and semiannual, active follow-up are based on postal questionnaires, with validation of reported events by the women's treating physicians. A multifaceted 4-level follow-up procedure will be established to ensure low loss to follow-up rates. The objective of the study is the investigation of the incidence of rare serious adverse events associated with the use of new and established OCs, and specifically the incidence of thromboembolic events.

DETAILED DESCRIPTION:
Active surveillance using valid epidemiologic study designs is desirable for any new product, because adverse effects may occur that have not yet been identified in pre-marketing studies.

The EURAS study investigates the safety of oral contraceptives with a large cohort of women attending offices of prescribing physicians. Its primary objective will be to compare incidence rates of adverse events in users of so-called new OCs and users of other OCs. The study is conducted as a phase IV commitment to the European Drug Authorities.

The combined cohort will include 50,000 to 60,000 women recruited by a selected set of physicians in six European countries. A total of more than 1,500,000 cycles are expected to be observed during the field work which will start early in 2001 and end early in 2006.

The participating women will undergo a baseline survey using a self administered questionnaire to describe the baseline risk. Every six months they will fill out a questionnaire in which they will record complaints and events during the use of the prescribed OC which will be validated. A multifaceted 4-level follow-up procedure will be established to ensure low loss to follow-up rates.

Based on experience obtained in previous OC studies complex sources of bias and confounding are expected. Thus, multivariate methods such as Cox regression will be used to adjust for confounding. Regarding the impact of the results on public health, the main emphasis will be on the absolute risk estimates.

ELIGIBILITY:
Inclusion Criteria:

* Women starting OC use or women switching OCs
* Women willing to participate in the active surveillance for several years

Exclusion Criteria:

* Women who have contraindications for OC use

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women prescribed hormonal contraceptives
Sampling Method: Non-Probability Sample
Enrollment: 59510 (Actual)
Dates: Start 2000-11; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Juergen C Dinger, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Result] Heinemann LA, Dinger J. Safety of a new oral contraceptive containing drospirenone. Drug Saf. 2004;27(13):1001-18. doi: 10.2165/00002018-200427130-00003. PMID 15471507
- [Result] Dinger JC, Heinemann LA, Kuhl-Habich D. The safety of a drospirenone-containing oral contraceptive: final results from the European Active Surveillance Study on oral contraceptives based on 142,475 women-years of observation. Contraception. 2007 May;75(5):344-54. doi: 10.1016/j.contraception.2006.12.019. Epub 2007 Feb 23. PMID 17434015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 59510 women were enrolled. Thereof 836 were excluded as they did not sign the informed consent form, were enrolled two or more times, continued their old OC or did not start OC use. In addition 371 used non oral hormonal contraception at study entry. These women were only used for the comparison of baseline risks.
Groups:
- Users of Drospirenone (DRSP): Women who use oral contraceptives (OCs) containing DRSP as progestin
- Users of Levonorgestrel (LNG): Women who use oral contraceptives (OCs) containing LNG as progestin
- Users of Other Oral Contraceptives (OCs): Women who use oral contraceptives (OCs) containing other progestins
Period: Overall Study
Arm/Group | Users of Drospirenone (DRSP) | Users of Levonorgestrel (LNG) | Users of Other Oral Contraceptives (OCs)
Started | 16534 | 15428 | 26341
Completed | 16133 (Numbers completed refer to first follow-up. Individual follow-up ranged between 1.5 and 5.0 years.) | 15009 (Numbers completed refer to first follow-up. Individual follow-up ranged between 1.5 and 5.0 years.) | 25762 (Numbers completed refer to first follow-up. Individual follow-up ranged between 1.5 and 5.0 years.)
Not Completed | 401 | 419 | 579

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Users of Drospirenone (DRSP) | Users of Levonorgestrel (LNG) | Users of Other Oral Contraceptives (OCs) | Total
Number analyzed (Participants) | 16534 | 15428 | 26341 | 58303
Age Categorical [Number; unit: participants]
  <=18 years | 3,454 | 4,215 | 6,307 | 13976
  Between 18 and 65 years | 13,080 | 11,213 | 20,034 | 44327
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.9 (8.1) | 25.1 (8.7) | 24.8 (7.8) | 25.2 (8.2)
Gender [Number; unit: participants]
  Female | 16,534 | 15,428 | 26,341 | 58303
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Europe | 16,534 | 15,428 | 26,341 | 58303

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolism (VTE)
Time Frame: 1.5 to 5 years
Population: The primary analysis compares the users of DRSP and LNG. Its results are presented below. The comparison of users of DRSP and OCs containing other progestins was only conducted for exploratory reasons. This secondary analysis showed similar results and is described in more detail in the publication of study results, see "citations".
Measure: Number; unit: Participants
Groups:
- Users of DRSP: Women who use authorized oral contraceptives containing DRSP prescribed by their gynecologist
- Users of LNG: Women who use authorized oral contraceptives containing LNG prescribed by their gynecologist
Arm/Group | Users of DRSP | Users of LNG
Number analyzed (Participants) | 16534 | 15428
Participants | 26 | 25
Statistical Analysis 1: Comparison: Users of DRSP vs Users of LNG; Null hypothesis: HR ≥ 2 (VTE of DRSP vs. LNG); Test type: Non-Inferiority or Equivalence — Sample size calculations for VTE risk showed that 50,000 patients should be sufficient to exclude a twofold risk; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.0, 95% CI [0.6 to 1.8]

ADVERSE EVENTS:
Time Frame: Between 1.5 and 5 years
Arm/Group | Users of Drospirenone (DRSP) | Users of Levonorgestrel (LNG) | Users of Other Oral Contraceptives (OCs)
Serious Adverse Events (participants affected / at risk) | 965/16534 | 1059/15428 | 1815/26341
Other Adverse Events (participants affected / at risk) | 0/16534 | 0/15428 | 0/26341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Users of Drospirenone (DRSP) (N=16534) | Users of Levonorgestrel (LNG) (N=15428) | Users of Other Oral Contraceptives (OCs) (N=26341)
Infectious diseases (Infections and infestations) | 51 | 48 | 82
Malignant neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 12 | 25
Benign neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 61 | 64 | 117
Diseases of the blood and blood-forming organs (Blood and lymphatic system disorders) | 3 | 3 | 12
Endocrine diseases (Endocrine disorders) | 34 | 47 | 55
Psychiatric and neurological diseases (Psychiatric disorders) | 43 | 58 | 109
Eye diseases (Eye disorders) | 10 | 17 | 27
Cardiovascular diseases (Cardiac disorders) | 91 | 99 | 171
Respiratory diseases (Respiratory, thoracic and mediastinal disorders) | 21 | 27 | 41
Digestive diseases (Gastrointestinal disorders) | 121 | 124 | 195
Skin diseases (Skin and subcutaneous tissue disorders) | 59 | 59 | 120
Diseases of the musculoskeletal system (Musculoskeletal and connective tissue disorders) | 151 | 162 | 261
Genitourinary diseases (Renal and urinary disorders) | 91 | 94 | 178
Injuries (Injury, poisoning and procedural complications) | 192 | 207 | 372
Other (General disorders) | 27 | 38 | 50

LIMITATIONS AND CAVEATS:
This is an observational study. The possibility of bias and residual confounding cannot be entirely eliminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes